CLINICAL TRIAL: NCT01958372
Title: Phase I Study of Thoracic Radiotherapy and Concurrent Chemotherapy With Soy Isoflavones in Stage III NSCLC (Non-Small Cell Lung Cancer) Patients
Brief Title: Radiation Therapy, Chemotherapy, and Soy Isoflavones in Treating Patients With Stage IIIA-IIIB Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gerold Bepler, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-021; NCI-2013-01835 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1307012220; 2013-021 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Bronchoalveolar Cell Lung Cancer; Large Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Soybean Proteins; Cisplatin; Etoposide; Pemetrexed; Radiotherapy

ARMS (2):
- Group I (squamous cell histology) (Experimental): Patients receive etoposide IV over 1 hour on days 1-5 and 29-33, cisplatin IV over 1 hour on days 1, 8, 29, and 36, and undergo RT 5 days a week for 6.6 weeks. Within 48 hours of initiating treatment, patients receive soy isoflavones PO daily on days 1-90.
  Interventions: Dietary Supplement: soy isoflavones; Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy
- Group II (non-squamous cell histology) (Experimental): Patients receive pemetrexed disodium IV over 10 minutes on days 1, 22, and 43 and cisplatin IV over 1 hour on days 1, 22, and 43. Patients also undergo RT and receive soy isoflavones as in Group I.
  Interventions: Dietary Supplement: soy isoflavones; Drug: cisplatin; Drug: pemetrexed disodium; Radiation: radiation therapy

INTERVENTIONS:
Dietary Supplement: soy isoflavones — Given PO
Drug: cisplatin — Given IV
Drug: etoposide — Given IV
  Arms: Group I (squamous cell histology)
Drug: pemetrexed disodium — Given IV
  Arms: Group II (non-squamous cell histology)
Radiation: radiation therapy — Undergo RT

SUMMARY:
This phase I trial studies the side effects of soy isoflavones when given together with radiation therapy and chemotherapy in treating patients with stage IIIA-IIIB non-small cell lung cancer. Radiation therapy uses high energy x rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, pemetrexed sodium, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Soy isoflavones may help radiation therapy, cisplatin, pemetrexed sodium, and etoposide work better by making tumor cells more sensitive to the drug. Soy isoflavones may also protect normal cells from the side effects of radiation therapy and chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of adding oral soy isoflavone to concurrent chemotherapy and radiotherapy for the treatment of patients with unresectable stage III non-small cell lung cancer (NSCLC).

OUTLINE: Patients are assigned to 1 of 2 treatment groups.

GROUP I (SQUAMOUS CELL HISTOLOGY): Patients receive etoposide intravenously (IV) over 1 hour on days 1-5 and 29-33, cisplatin IV over 1 hour on days 1, 8, 29, and 36, and undergo radiation therapy (RT) 5 days a week for 6.6 weeks. Within 48 hours of initiating treatment, patients receive soy isoflavones orally (PO) daily on days 1-90.

GROUP II (NON-SQUAMOUS CELL HISTOLOGY): Patients receive pemetrexed disodium IV over 10 minutes on days 1, 22, and 43 and cisplatin IV over 1 hour on days 1, 22, and 43. Patients also undergo RT and receive soy isoflavones as in Group I.

After completion of study treatment, patients are followed up at 4 weeks and then every 4 months for 1 year, every 6 months for 1 year, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of stage III non-small cell lung cancer; patients will need to meet the following criteria for stage IIIA or IIIB diagnosis:

  * IIIA

    * Histologic or cytologic diagnosis of ipsilateral mediastinal lymph node involvement, or
    * Tumors greater than 7 cm or with chest wall invasion, or involvement of one of the following diaphragm, phrenic nerve, mediastinal pleura or parietal pericardium with hilar or mediastinal lymph node involvement
    * More than one mediastinal lymph node enlarged on computed tomography (CT) scan and the same lymph nodes positive on positron emission tomography (PET) scans or
    * Paralyzed left vocal cord with separate lung primary distinct from the aorto-pulmonary lymph nodes on the CT scan
  * IIIB

    * Histologic or cytologic diagnosis of N3 lymph node involvement; or
    * Enlarged N3 lymph nodes on CT scan that are positive on PET scan as well; patient must not have extension of lymph node involvement to cervical lymph nodes other than supraclavicular lymph nodes; or
    * Right sided primary with left vocal cord paralysis; or
    * Evidence of tumor extension into the mediastinum and/or mediastinal structures either at the time of mediastinoscopy, bronchoscopy or on CT scans
    * Patients with a nodules in the same lung but no other areas of involvement
    * Patients with prior surgically resected stage I NSCLC who did not receive any adjuvant therapy, who now have stage IIIA or B NSCLC will be eligible
* Southwestern Oncology Group (SWOG) performance status 0 or 1
* Absolute neutrophil count of > 1.5 x 10^9/L
* Platelet count > 100,000 x 10^9/L
* Serum creatinine =< 1.5 times the institutional upper limit of normal (ULN)
* Calculated creatinine clearance (Cockcroft-Gault formula) of >= 45mL/min
* Serum bilirubin > ULN
* Transaminases (serum glutamic oxaloacetic transaminase [SGOT] and/or serum glutamate pyruvate transaminase [SGPT]) > 1.5 times institutional ULN
* Alkaline phosphatase >= 2.5 times ULN
* Forced expiratory volume in one second (FEV1) of >= 1 liter and diffusion capacity of carbon monoxide (DLCO) >= 40% of predicted
* Patient should undergo brain imaging (CT scan or magnetic resonance imaging [MRI ]) to rule out brain metastases
* Signed informed consent that details the investigational nature of the study according to institutional and federal guidelines
* Registered with Clinical Trials Office at Karmanos Cancer Institute/Wayne State University

Exclusion Criteria:

* Prior chemotherapy, radiation for any malignancy in which they received any thoracic radiotherapy
* Patients with concurrent malignancy; patients with prior or concurrent malignancy will be allowed as long as the treating physician considers it unlikely to impact the clinical outcome of the patient
* Patients with peripheral neuropathy > 2
* Serious medical illness including but not limited to uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction or cerebrovascular event with 6 months of registration, history of chronic active hepatitis or history of human immunodeficiency virus (HIV) or an active bacterial infection will not be eligible
* Inability or unwillingness to take folic acid or vitamin B12 or dexamethasone
* Pregnant or lactating women; all pre-menopausal and peri-menopausal women should have a urine test for pregnancy within a week of starting therapy; all patients of child bearing potential should agree to use an effective contraceptive method
* Patients should not participate in any other therapeutic investigational study while taking part in this study
* Patients on warfarin will not be allowed on the study; patient on low molecular heparin or anti direct factor Xa inhibitor (Xa) drugs will be allowed
* Patients with a soy allergy will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-08; Primary Completion 2017-10-09 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Safety, in terms of dose-limiting toxicity of adding oral soy isoflavone supplementation to concurrent chemotherapy and radiotherapy, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 | Up to 90 days
Survival proportion | 1 year

SECONDARY OUTCOMES:
Grade 3-4 toxicity rate graded according to NCI CTCAE version 4.0 | Up to 2 years
  Point and exact confidence interval estimates of the grade 3-4 toxicity rate will be computed for each type of toxicity encountered.
Response (complete response [CR] and partial response [PR]) rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 2 years
  Point and exact confidence interval estimates of the (complete + partial) response rate will be computed.
Time to tumor progression (TTP) | From the date of registration until the date that PD (progressive disease) or death is first reported, assessed up to 2 years
  TTP will be estimated using standard Kaplan-Meier methods for censored data, from which the median and other statistics of interest will be calculated (e.g., rates at 3 months, 6 months, 12 months).
Overall survival (OS) | From the date of registration to the date of death, assessed up to 2 years
  OS will be estimated using standard Kaplan-Meier methods for censored data, from which the median and other statistics of interest will be calculated (e.g., rates at 3 months, 6 months, 12 months).
Response duration | From the time that measurement criteria are first met for CR until the date that PD is objectively documented, assessed up to 2 years
  Response duration will be estimated using standard Kaplan-Meier methods for censored data, from which the median and other statistics of interest will be calculated (e.g., rates at 3 months, 6 months, 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Shirish Gadgeel, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (5):
- United States (5):
  - Karmanos Cancer Institute at McLaren Bay Region, Bay City, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute at McLaren Lapeer Region, Lapeer, Michigan
  - Karmanos Cancer Institute at McLaren Central Michigan, Mount Pleasant, Michigan
  - Karmanos Cancer Institute at McLaren Northern, Petoskey, Michigan